CLINICAL TRIAL: NCT01444222
Title: Behaviour of Tricuspid Valve Regurgitation in Volume and/or Pressure Loaded Right Heart
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s53471
Record Dates: First submitted 2011-09-27; First posted 2011-09-30 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2011-01

CONDITIONS: Tricuspid Valve Insufficiency
Keywords: Myocardial contractility; Quantification of regurgitant flow; exercise capacity
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Pulmonary Hypertension
- pulmonic valve stenosis
- pulmonic valve homograft
- pulmonic valve insufficiency
- atrial septum defect
- Ebstein's anomaly
- transvalvular right ventricular lead
- control

SUMMARY:
Right-sided heart disease has an important impact on the prognosis of patients with valvular heart disease. Up to now, Tricuspid Valve Regurgitation (TR) and right heart hemodynamics have not been extensively investigated. However, it is plausible that a significant degree of TR and the associated volume-overload of the right ventricle cause significant right ventricular wall stress. Although minor TR generally is well tolerated, major TR can lead to clinical symptoms, right ventricular dilatation and ultimately right ventricular heart failure. Up to now, the investigators do not dispose of any tools to diagnose and anticipate this unfavourable evolution. Nevertheless it is likely that right ventricular failure is preceded with a subclinical dysfunction of the right ventricle and a possibly reversible change in contractility of the myocardium.

Recently, new techniques to evaluate the systolic function, the contractility and the hemodynamics of the heart have become available.

First, this study will help us assessing the feasibility and accuracy of several imaging modalities in right-sided heart pathology with focus on TR and right heart myocardial performance.

Second, this study will contribute to a better understanding of the hemodynamic effect of volume-overload and/or pressure-overload of the right ventricle. It will clarify the behaviour of TR, the evolution of right ventricular myocardial contractility and dysfunction during exercise and its impact on exercise capacity. By doing this, discrimination between well tolerated and ill-tolerated TR will be possible, thus identifying patients who might be eligible for treatment (medical, corrective, …).

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary Arterial Hypertension
* Pulmonic Valve Stenosis
* Pulmonic valve homograft
* Pulmonic valve insufficiency
* Atrium Septum Defect
* Ebstein's Anomaly
* Transvalvular RV pacemaker/ shock lead
* Control

Exclusion Criteria:

* age < 16 years
* not fit for bicycle testing

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Pulmonary Arterial Hypertension
  * Pulmonic Valve Stenosis
  * Pulmonic valve insufficiency
  * Atrium Septum Defect
  * Ebstein's Anomaly
  * Transvalvular RV pacemaker/ shock lead
  * Control
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-10-18 (Actual); Primary Completion 2013-05-24 (Actual); Study Completion 2014-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Budts, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] De Meester P, Buys R, Van De Bruaene A, Gabriels C, Voigt JU, Vanhees L, Herijgers P, Troost E, Budts W. Functional and haemodynamic assessment of mild-to-moderate pulmonary valve stenosis at rest and during exercise. Heart. 2014 Sep;100(17):1354-9. doi: 10.1136/heartjnl-2014-305627. Epub 2014 Apr 29. PMID 24780907